CLINICAL TRIAL: NCT06387108
Title: Evaluation of a Training Course for Educational Professionals on Depression and Mental Health in Childhood and Adolescence
Brief Title: Evaluation of a Training Course for Educational Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Lisa Feldmann, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-0045
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Depression; Depression in Children; Depression in Adolescence
Keywords: Knowledge; Mental Health; Depression Literacy; Training course; Educational professionals; School intervention; Evaluation
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2 hours online training (Experimental): 2 hours online training for educational professionals about depression and mental health in youths
  Interventions: Other: training course

INTERVENTIONS:
Other: training course — Two-hour online training course for educational professionals at schools on depression and mental health in children and adolescents (including symptoms, causes, comorbidity, prevention) and practical tips for everyday school life to reduce stress.

SUMMARY:
The aim of this study is to evaluate the efficacy of a two-hour online training course on depression and mental health in childhood and adolescence in educational professionals to improve depression and mental health literacy. It will further be investigated whether the course leads to changes in attitudes towards the illness (reduction of stigma) and to an increased behavioural confidence and behavioral change in dealing with pupils with symptoms and illnesses.

DETAILED DESCRIPTION:
Depressive disorders are among the most common psychiatric disorders in childhood and adolescence and yet often are unnoticed and not treated for a long time. Depressive disorders often begin in adolescence and young adulthood. School stress, caused by bullying experiences at school or high performance expectations from parents and teachers, has been identified as an important factor in the development of depressive disorders in students School, as a central area of life for children and young people, is an important place for promoting pupils' mental health.

The rising prevalence of depressive disorders among adolescence in recent years and the delayed start of interventions show a clear need for action in the everyday lives of adolescents. A training for educational professionals in schools on depression in youths is intended to reduce the large treatment gap. By educating about depression, reducing stigma and fostering confidence in dealing with pupils with depression, educational professionals at schools should be sensitised to youth depression so that they can better respond to pupils with mental health problems.

As part of the planned scientific study, a training course on depression and mental health in childhood and adolescence for educational professionals is to be evaluated. The study will investigate the extent to which a two-hour online training course on depression and mental health in childhood and adolescence (including symptoms, causes of depression, comorbid diseases, prevention) and practical tips for everyday school life leads to an increase in knowledge regarding these topics. Additionally, the study will investigate the impact of the training on changes in attitudes towards depression (reduction of stigma), increased behavioural confidence dealing with pupils with mental health problems and changes in behavior deadling pupils with mental health problems. Moreover, the influence of teachers' emotions (assessed via the Teachers Emotion Scales) and self-efficacy on the outcomes will be exploratively investigated. To this end, the educational professionals will take part in 3 online surveys (before the training, shortly after the training and 4 weeks after the training) via Limesurvey.

ELIGIBILITY:
Inclusion Criteria:

* Current teaching profession (teacher) / working in the school environment (e.g. school psychologist, social worker)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
increase in Knowledge | pre (0-1 days before the training), post (0-1 days after training) and 1month follow-up
  Self-designed questionnaire based on the 2 hours depression and mental health training
decrease in depression stigma | pre (0-1 days before the training), post (0-1 days after training) and 1month follow-up
  Assessed via Depression Stigma Scale (DSS, Griffiths, Christensen, & Jorm, 2008)

SECONDARY OUTCOMES:
Change in helping behaviour towards pupil | pre (0-1 days before the training), 1month follow-up
  Self-designed questionnaire based on Jorm, Kitchener, Sawyer, Scales, & Cvetkovski, 2010; Parker et al., 2021; Sebbens, Hassmén, Crisp, & Wensley, 2016
Change in conficende in dealing with pupils with mental health issues | pre (0-1 days before the training), post (0-1 days after training) and 1month follow-up
  self-designed questionnaire based on Sebbens, 2016; Parker, 2021

OTHER OUTCOMES:
Evaluation of the training | post (0-1 days after training)
  Self-designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital
Locations (1):
- LMU University Hospital (recruitment is conducted online), Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths KM, Christensen H, Jorm AF. Predictors of depression stigma. BMC Psychiatry. 2008 Apr 18;8:25. doi: 10.1186/1471-244X-8-25. PMID 18423003
- [Background] Jorm AF, Kitchener BA, Sawyer MG, Scales H, Cvetkovski S. Mental health first aid training for high school teachers: a cluster randomized trial. BMC Psychiatry. 2010 Jun 24;10:51. doi: 10.1186/1471-244X-10-51. PMID 20576158
- [Background] Parker BL, Anderson M, Batterham PJ, Gayed A, Subotic-Kerry M, Achilles MR, Chakouch C, Werner-Seidler A, Whitton AE, O'Dea B. Examining the Preliminary Effectiveness and Acceptability of a Web-Based Training Program for Australian Secondary School Teachers: Pilot Study of the BEAM (Building Educators' Skills in Adolescent Mental Health) Program. JMIR Ment Health. 2021 Oct 22;8(10):e29989. doi: 10.2196/29989. PMID 34677134
- [Background] Sebbens J, Hassmen P, Crisp D, Wensley K. Mental Health in Sport (MHS): Improving the Early Intervention Knowledge and Confidence of Elite Sport Staff. Front Psychol. 2016 Jun 24;7:911. doi: 10.3389/fpsyg.2016.00911. eCollection 2016. PMID 27445887
- [Background] Schwarzer, R., & Jerusalem, M. (2003). SWE. Skala zur Allgemeinen Selbstwirksamkeitserwartung [Verfahrensdokumentation, Autorenbeschreibung und Fragebogen]. In L.-I. f. P. (ZPID) (Ed.), Open Test Archive. Trier: ZPID.
- [Background] Frenzel, A. C., Pekrun, R., Goetz, T., Daniels, L. M., Durksen, T. L., Becker-Kurz, B., & Klassen, R. M. (2016). Measuring Teachers' enjoyment, anger, and anxiety: The teacher emotions scales (TES). Contemporary Educational Psychology, 46, 148-163.
- [Background] Sacco R, Camilleri N, Eberhardt J, Umla-Runge K, Newbury-Birch D. A systematic review and meta-analysis on the prevalence of mental disorders among children and adolescents in Europe. Eur Child Adolesc Psychiatry. 2024 Sep;33(9):2877-2894. doi: 10.1007/s00787-022-02131-2. Epub 2022 Dec 30. PMID 36581685
- [Background] Soneson, E., & Ford, T. (2020). Identifying mental health difficulties in children & young people: the role of schools - ACAMH, The Association for Child an Adolescent Mental Health. doi:10.13056/acamh.13021
- [Background] Solmi M, Radua J, Olivola M, Croce E, Soardo L, Salazar de Pablo G, Il Shin J, Kirkbride JB, Jones P, Kim JH, Kim JY, Carvalho AF, Seeman MV, Correll CU, Fusar-Poli P. Age at onset of mental disorders worldwide: large-scale meta-analysis of 192 epidemiological studies. Mol Psychiatry. 2022 Jan;27(1):281-295. doi: 10.1038/s41380-021-01161-7. Epub 2021 Jun 2. PMID 34079068
- [Background] Li W, Zhao Z, Chen D, Peng Y, Lu Z. Prevalence and associated factors of depression and anxiety symptoms among college students: a systematic review and meta-analysis. J Child Psychol Psychiatry. 2022 Nov;63(11):1222-1230. doi: 10.1111/jcpp.13606. Epub 2022 Mar 16. PMID 35297041
- [Background] Schulte-Körne, G. (2016). Psychische Störungen bei Kindern und Jugendlichen im schulischen Umfeld. 113(11), 183-190. doi:10.3238/arztebl.2016.0183
- [Background] Ye Z, Wu D, He X, Ma Q, Peng J, Mao G, Feng L, Tong Y. Meta-analysis of the relationship between bullying and depressive symptoms in children and adolescents. BMC Psychiatry. 2023 Mar 30;23(1):215. doi: 10.1186/s12888-023-04681-4. PMID 36997959
- [Background] Tong Y, Wang S, Cao L, Zhu D, Wang F, Xie F, Zhang X, Wang G, Su P. School dropouts related to mental disorders: A systematic review and meta-analysis. Asian J Psychiatr. 2023 Jul;85:103622. doi: 10.1016/j.ajp.2023.103622. Epub 2023 May 8. No abstract available. PMID 37172421
- [Background] Doll CM, Michel C, Rosen M, Osman N, Schimmelmann BG, Schultze-Lutter F. Predictors of help-seeking behaviour in people with mental health problems: a 3-year prospective community study. BMC Psychiatry. 2021 Sep 3;21(1):432. doi: 10.1186/s12888-021-03435-4. PMID 34479537
- [Background] Thapar A, Eyre O, Patel V, Brent D. Depression in young people. Lancet. 2022 Aug 20;400(10352):617-631. doi: 10.1016/S0140-6736(22)01012-1. Epub 2022 Aug 5. PMID 35940184
- [Background] Liao Y, Ameyaw MA, Liang C, Li W. Research on the Effect of Evidence-Based Intervention on Improving Students' Mental Health Literacy Led by Ordinary Teachers: A Meta-Analysis. Int J Environ Res Public Health. 2023 Jan 4;20(2):949. doi: 10.3390/ijerph20020949. PMID 36673704
- [Background] Coppens E, Van Audenhove C, Iddi S, Arensman E, Gottlebe K, Koburger N, Coffey C, Gusmao R, Quintao S, Costa S, Szekely A, Hegerl U. Effectiveness of community facilitator training in improving knowledge, attitudes, and confidence in relation to depression and suicidal behavior: results of the OSPI-Europe intervention in four European countries. J Affect Disord. 2014 Aug;165:142-50. doi: 10.1016/j.jad.2014.04.052. Epub 2014 May 4. PMID 24882192
- [Background] Vieira MA, Gadelha AA, Moriyama TS, Bressan RA, Bordin IA. Evaluating the effectiveness of a training program that builds teachers' capability to identify and appropriately refer middle and high school students with mental health problems in Brazil: an exploratory study. BMC Public Health. 2014 Feb 28;14:210. doi: 10.1186/1471-2458-14-210. PMID 24580750
- [Background] Danielsen, A. G., Samdal, O., Hetland, J., & Wold, B. (2009). School-related social support and students' perceived life satisfaction. The Journal of Educational Research, 102(4), 303-318. doi:10.3200/JOER.102.4.303-320
- [Background] Jiang, X., Huebner, E. S., & Siddall, J. (2013). A Short-Term Longitudinal Study of Differential Sources of School-Related Social Support and Adolescents' School Satisfaction. Social Indicators Research, 114(3), 1073-1086. doi:10.1007/s11205-012-0190-x
- [Background] Plenty S, Ostberg V, Almquist YB, Augustine L, Modin B. Psychosocial working conditions: an analysis of emotional symptoms and conduct problems amongst adolescent students. J Adolesc. 2014 Jun;37(4):407-17. doi: 10.1016/j.adolescence.2014.03.008. Epub 2014 Mar 31. PMID 24793388
- [Background] Pullmann, M., Bruns, E., Daly, B., & Sander, M. (2013). Improving the evaluation and impact of mental health and other supportive school-based programmes on students' academic outcomes. Advances in School Mental Health Promotion, 6, 226-230. doi:10.1080/1754730x.2013.835543
- [Background] Weist MD, Hoover SA, Daly BP, Short KH, Bruns EJ. Propelling the Global Advancement of School Mental Health. Clin Child Fam Psychol Rev. 2023 Dec;26(4):851-864. doi: 10.1007/s10567-023-00434-7. Epub 2023 May 29. PMID 37247024
- [Derived] Saffenreuther AK, Greimel E, Primbs R, Iglhaut L, Kaubisch S, Schulte-Korne G, Feldmann L. Evaluation of an online training course for educational professionals on depression and mental health in childhood and adolescence. Child Adolesc Psychiatry Ment Health. 2025 Dec 15. doi: 10.1186/s13034-025-01007-y. Online ahead of print. PMID 41398959